CLINICAL TRIAL: NCT01427218
Title: A Prospective Evaluation of a Medication Therapy Management Clinic Versus Usual Medical Care in Patients Post Acute Coronary Syndrome: The MUMPS Study
Brief Title: Monitoring and Adjustment of Medication Therapy for Patients With Heart Disease
Acronym: MUMPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Middle Tennessee Research Institute (Other)
Collaborators: American Society of Health-System Pharmacists Research and Education Foundation (Other)
Responsible Party: Principal Investigator, James A S Muldowney, III MD, Assistant Professor of Medicine, Vanderbilt Univ. School of Med, Middle Tennessee Research Institute
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2010100590
Record Dates: First submitted 2011-01-14; First posted 2011-09-01 (Estimated); Last update posted 2011-09-01 (Estimated); Status verified 2011-08

CONDITIONS: Coronary Heart Disease; Myocardial Infarction
Keywords: pharmacist; medication therapy management; evidence based medicine
MeSH Terms: conditions — Coronary Disease; Myocardial Infarction | interventions — Medication Therapy Management; Medication Reconciliation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medication Therapy Management (MTM) (Experimental): Medication Therapy Management visits with a pharmacotherapist will occur at a minimum of 6-9 weeks, 20-24 weeks, and 28-32 weeks. Additional interim face to face and telephonic visits may be scheduled based on patient's progress with meeting treatment goals and need for follow-up physical assessment and laboratory analysis.
  Interventions: Other: Titration of medications; Behavioral: Lifestyle Counseling; Behavioral: Medication Counseling
- Usual Care (Placebo Comparator): Visits with a pharmacotherapist to create an accurate list of medications for those patients randomized to placebo (who receive usual care by their cardiologist and primary care provider).
  Interventions: Other: Usual Care with Medication Reconciliation

INTERVENTIONS:
Other: Titration of medications — Titration of medications for cholesterol, blood pressure, heart failure, and angina will occur. Cholesterol medications will be titrated according to labs at intervals nor more frequently than every 6 weeks until target LDL reached. Blood pressure (BP) medications will be titrated no more frequently than every 1-2 weeks until target BP reached. Heart failure medications will be titrated no more frequently than every 1-2 weeks until target doses reached or clinical status goals achieved. Anginal (chest pain) medications will be titrated no more frequently than every 1-2 weeks until control of chest pain occurs. Some patients will require more titrations than other patients (titration is patient specific).
  Other Names: Medication Therapy Management
  Arms: Medication Therapy Management (MTM)
Behavioral: Lifestyle Counseling — The pharmacist will provide counseling on diet modification, smoking cessation, and physical activity
  Other Names: Medication Therapy Management
  Arms: Medication Therapy Management (MTM)
Behavioral: Medication Counseling — The pharmacist will counsel the patient on adherence aids and medication safety and efficacy self and clinical monitoring.
  Other Names: Medication Therapy Management
  Arms: Medication Therapy Management (MTM)
Other: Usual Care with Medication Reconciliation — A medication history and assessment of adherence will be completed by the pharmacist.
  Other Names: Usual Physician Care
  Arms: Usual Care

SUMMARY:
Existing trials for the patient with coronary heart disease evaluate the interdisciplinary team dynamic where pharmacists (pharmacotherapists) provide therapeutic recommendations in the inpatient environment. To our knowledge, only other trial has evaluated the addition of a pharmacist (or nurse practitioner) in an outpatient collaborative cardiology practice and has found no benefit. However, the investigators believe that since a cardiology based pharmacist (pharmacotherapist) in the Veterans Health Administration has physical assessment skills, a shorter cycle length between appointments, and the ability to provide medication therapy management, the pharmacotherapist should be similarly successful as seen with other pharmacist based medication therapy management practices. The investigators will assess effectiveness by using the combined endpoint of blood pressure and lipid treatment. Additionally the investigators will conduct three substudies to evaluate if the pharmacist can improve all cause mortality and cardiovascular morbidity, adherence to antihypertensives, and patient satisfaction.

DETAILED DESCRIPTION:
Existing trials for the patient with coronary heart disease evaluate the interdisciplinary team dynamic where pharmacists (pharmacotherapists) provide therapeutic recommendations in the inpatient environment. To our knowledge, only other trial has evaluated the addition of a pharmacist (or nurse practitioner) in an outpatient collaborative cardiology practice and has found no benefit. However, the investigators believe that since a cardiology based pharmacist (pharmacotherapist) in the Veterans Health Administration has physical assessment skills, a shorter cycle length between appointments, and the ability to provide medication therapy management, the pharmacotherapist should be similarly successful as seen with other pharmacist based medication therapy management practices. The investigators will assess effectiveness by using the combined endpoint of blood pressure and lipid treatment. Additionally the investigators will conduct three substudies to evaluate if the pharmacist can improve all cause mortality and cardiovascular morbidity, adherence to antihypertensives, and patient satisfaction.

This is a randomized study comparing the use of a medication therapy management clinic improves cardiac risk factors and recurrent hospitalization in patients admitted with an acute coronary syndrome.

100 subjects will be enrolled as a minimum. Patients will be randomized to usual care or enrollment in the MTM clinic where they will be seen every two months for 8 months.

The primary endpoint is blood pressure and lipid changes. Secondary endpoints include satisfaction with pharmacists, medication habit changes, recurrent events.

ELIGIBILITY:
Inclusion Criteria:

All patients with a diagnosis of ACS at the VA Tennessee Valley Healthcare System who

1. are greater than or equal to 60 years of age
2. will benefit from Medication Therapy Management (MTM):

   * Have a baseline LDL >79mg/dL in the first 24 hours of acute coronary syndrome (ACS) OR if LDL not assessed in the first 24 hours of ACS, have a recent LDL >79mg/dL (in the last 15 months) OR not have an LDL assessed prior to or during admission.

   AND
   * Have outpatient blood pressures (BP) above goal on 65% or more of assessments within the last 15 months or a SBP >140mmHg or DBP>90mmHg or both on the last outpatient BP assessment.
3. are enrolled or will be enrolled in outpatient cardiovascular services at the VA Tennessee Valley Healthcare System

Exclusion Criteria:

Patients who

1. are transferred to a long-term care facility or skilled nursing facility
2. are assigned to another Veterans Health Administration medical center,
3. have a discharge primary or secondary discharge diagnosis code for dementia, schizophrenia, or organic brain syndrome,
4. cannot speak or understand English or give written informed consent,
5. are enrolled in hospice or palliative care
6. are participating in another trial that prohibits participation in this trial
7. have a baseline LDL> 200mg/dL in proximity to admission suggestive of familial hypercholesterolemia (FH) or a known diagnosis of FH
8. require clonidine or minoxidil for blood pressure control prior to the index admission
9. are enrolled in the Nashville preventative cardiovascular clinic for hypertension
10. have a urinary drug screen positive for cocaine in the last 12 months
11. have plans to move in the next 6 months

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2010-11; Primary Completion 2012-09 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients at guideline goal for both blood pressure and lipids | 28-32 weeks after enrollment (final study visit)
  The Primary endpoint is the percentage of patients in each group who have BOTH their lipids AND their BP controlled within guideline specifications at the end of the study in order to determine if the clinic improves control of BOTH of these risk factors. (e.g. on the final study visit, 75% in the intervention arm and 50% in the control arm have controlled lipids AND blood pressure, given the I/E criteria, both groups start out at 0% at entry).

SECONDARY OUTCOMES:
Composite cardiovascular morbidity and all-cause mortality | 6-9 weeks and 28-32 weeks after enrollment
  A between group comparison of all cause mortality or VA cardiovascular readmission.
Patient Satisfaction with Clinical Pharmacist Services | 28-32 weeks
  A descriptive analysis to assess patients' feelings about the pharmacist being involved in their CHD care
Change in Adherence with 8-item Morisky Adherence Tool | 6-9 weeks and 28-32 weeks
  A within group comparison of the adherence score to determine if the relationship with the pharmacist may assist with (subjective) adherence with antihypertensive therapy.

CONTACTS AND LOCATIONS:
Overall Officials: James AS Muldowney, III, MD, Principal Investigator — VA Tennessee Valley Healthcare System
Locations (1):
- VA Tennessee Valley Healthcare System, Nashville, Tennessee, United States